CLINICAL TRIAL: NCT04005586
Title: A Prospective Controlled Multi-Center Clinical Study to Evaluate The Safety and Effectiveness of Performing 0.50 Diopter Astigmatism Correction on the Commercially Available RxSight Light Adjustable Lens (LAL)
Brief Title: A Clinical Study to Evaluate The Safety and Effectiveness of Performing 0.50 Diopter Astigmatism Correction on the Commercially Available RxSight Light Adjustable Lens (LAL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RxSight, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP-034
Record Dates: First submitted 2019-06-26; First posted 2019-07-02 (Actual); Results first posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Aphakia; Cataract
Keywords: Light Delivery Device; LDD; Intraocular lens; Light Adjustable Lens; LAL
MeSH Terms: conditions — Aphakia; Cataract

STUDY DESIGN:
Intervention Model Description: All subjects will receive the same treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Light Delivery Device (LDD) (Experimental): Patient's study eye will undergo light delivery treatments to the commercially available light adjustable lens.
  Interventions: Device: Light Delivery Device (LDD)

INTERVENTIONS:
Device: Light Delivery Device (LDD) — Study eye will undergo Light delivery Device treatments

SUMMARY:
The primary objective of this study is to evaluate the safety and effectiveness of performing 0.50 D cylinder correction on the RxSight Light Adjustable Lens (LAL) in patients who have undergone implantation with the FDA approved, commercially available LAL.

ELIGIBILITY:
Inclusion Criteria:

* A study eye implanted with the commercially approved LAL that has not undergone any previous LDD treatments
* A study eye with manifest refraction cylinder of 0.50 D measured by two independent examiners at the Adjustment #1 visit prior to the first light adjustment treatment.
* Sign a written Informed Consent form and be willing to receive light treatment for their 0.50 D of cylinder.
* Between the ages of 40 and 80 inclusive on the day the informed consent form is signed.
* Good vision in the fellow eye with best corrected distance visual acuity (BCDVA) 20/40 or better.
* Willing and able to comply with the requirements for study specific procedures and visits

Exclusion Criteria:

* Pre-existing macular disease in the study eye.
* History of uveitis in the study eye.
* Has undergone previous corneal or intraocular surgery in the study eye, except for the cataract surgery and eyes with previous pterygium excision are permitted as long as the pterygium did not extend more than 2mm onto the cornea from the limbus.
* Subjects taking systemic medication that may increase sensitivity to UV light.
* Subjects taking a systemic medication that is considered toxic to the retina such as tamoxifen.
* History of ocular herpes simplex virus in the study eye.
* Subject who has participated within another ophthalmic clinical trial within the last 3 months.
* Sutures used at the time of surgery to close the incision wound in the study eye

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cleveland Eye Clinic, Brecksville, Ohio
  - Vance Thompson Vision Clinic, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Light Delivery Device (LDD)
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Light Delivery Device (LDD)
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | NA — Data not collected
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Mean Manifest Refraction Cylinder (MRCYL) Compared Between the Three Study Groups, LAL Treatment Group and Historical Control Groups
Time Frame: Post Op Month 3
Measure: Mean (Standard Deviation); unit: Diopter (D)
Arm/Group | Light Delivery Device (LDD)
Number analyzed (Participants) | 25
Diopter (D) | -0.14 (0.21)
Statistical Analysis 1: Comparison: Light Delivery Device (LDD); Two different historical controls implanted under NCT01496066 were used; Test type: Other — The comparison was made by descriptive statistics; The LAL treatment group had a mean MRCYL of -0.14 (+/- 0.21D) compared to -0.33 (+/- 0.29D) and -0.40 (+/- 0.36D) for the LAL historical control group and the monofocal IOL historical control group in NCT01496066 respectively

2. Primary Outcome: Change in Manifest Refraction Cylinder (MRCYL) Compared Between the Three Study Groups, LAL Treatment Group and Historical Control Groups
Time Frame: Post Op Month 3
Measure: Mean (Standard Deviation); unit: Diopter (D)
Arm/Group | Light Delivery Device (LDD)
Number analyzed (Participants) | 25
Diopter (D) | 0.36 (0.21)
Statistical Analysis 1: Comparison: Light Delivery Device (LDD); Two different historical controls implanted under NCT01496066 were used; Test type: Other — The comparison was made by descriptive statistics; The LAL treatment group MRCYL change from baseline was 0.36 (+/- 0.21D) compared to 0.17 (+/- 0.29D) and 0.10 (+/- 0.36D) for the LAL historical control group and the monofocal IOL historical control group in NCT01496066, respectively

3. Other Pre Specified Outcome: Safety: ISO 11979-7 Number of Eyes With Ocular Adverse Events (Device Related and Unrelated)
Description: Number of study eyes experiencing Ocular adverse events (device related and unrelated)
Time Frame: Through study completion, an average of 3 months
Population: Safety population
Measure: Number; unit: eyes
Arm/Group | Light Delivery Device (LDD)
Number analyzed (Participants) | 25
eyes | 4

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 3 months.
Description: Non-ocular adverse events were not collected. Adverse events were counted by eye.
Arm/Group | Light Delivery Device (LDD)
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 4/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Light Delivery Device (LDD) (N=25)
Non-clinically significant cystoid macular edema (Eye disorders) | 1 (1)
Non-clinically significant cystoid macular edema in non-study eye (Eye disorders) | 1 (1)
Posterior Capsular Opacity (PCO) that requires YAG Capsulotomy treatment (Eye disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-23): https://cdn.clinicaltrials.gov/large-docs/86/NCT04005586/Prot_SAP_000.pdf